CLINICAL TRIAL: NCT01376596
Title: Manualized Group Cognitive-behavioral Intervention for Social Anxiety in Schizophrenia: An Efficacy Pilot Study.
Brief Title: Group Cognitive-behavioral Intervention for Social Anxiety in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Martin Lepage, Psychiatry professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-273-PSY
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Social Anxiety; Schizophrenia
Keywords: Remission; Psychosocial Functioning; Symptoms reduction
MeSH Terms: conditions — Schizophrenia | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-based Intervention (Experimental): Contrast the impact of a CBT intervention for the treatment of social anxiety in schizophrenia with standard care (care as usual)
  Interventions: Behavioral: Cognitive-Behavioral Therapy based intervention immediately
- Treatment as usual (Active Comparator): Usual care received by patients at clinic/hospital - randomized to a wait list to receive the CBT intervention at the end of the group that received the intervention immediately
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy based intervention immediately — This intervention will include: i) Psychoeducation on social anxiety disorder; ii) Cognitive Restructuring: Identify negative thoughts that occur before, during, or after anxiety-provoking situations; Evaluate the accuracy of their thoughts in the light of data derived from Socratic questioning or as a result of so-called behavioral experiments; and derive rational alternative thoughts based on the acquired information; iii) Exposure component, which focuses on the collection of information that will allow patients to revise their judgments about the degree of risk to which they are exposed in feared situations, challenge their dysfunctional beliefs about the self relative to the illness and their self-efficacy (social status related), and iv) Use of Thought Records to identify, explore and dispute negative thoughts about dysfunctional self-identity and core beliefs related to the onset and presence of diagnosis of schizophrenia.
  Arms: CBT-based Intervention
Behavioral: Wait list — The group receiving treatment as usual (TAU) will be put on a wait list to receive the CBT intervention at the end of the experimental group, the one receiving the intervention immediately
  Arms: Treatment as usual

SUMMARY:
This study will explore the helpfulness of a short psychological group treatment called cognitive-behavioral therapy, or CBT. CBT is a form of therapy that is very structured and it aims to improve difficulties that are related to behaviors and emotions by first working on identifying and changing negative inaccurate thoughts. The main goal of this intervention is to see if group CBT reduces the symptoms of social anxiety in people with schizophrenia so that they can improve their social functioning and help their psychotic symptoms. The study compares the usefulness of adding CBT to standard services.

DETAILED DESCRIPTION:
Social anxiety is highly prevalent in people with schizophrenia and represents a major obstacle to positive functional outcomes. Social anxiety is a treatable condition but has, in the context of psychosis, received only scant attention thus far. Current existing manualized treatment for social anxiety may not be optimal for people with schizophrenia for a number of reasons described above. An adapted CBT intervention for schizophrenia must target the stigma attached to the illness, the presence of poor social skills, the presence of delusional and persecutory ideas, possible limited reading abilities, and associated cognitive deficits. The investigators propose to develop and test an adapted group CBT for social anxiety. The main objective of this research proposal is to contrast the impact of a CBT intervention for the treatment of social anxiety in schizophrenia with standard care (care as usual) on reducing symptoms of social anxiety. Considering the relationship between certain characteristics of social anxiety (e.g. social withdrawal) with diminished quality of life and poor functional outcome, a secondary objective is to examine the impact of reduced social anxiety on functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a schizophrenia spectrum disorder; aged 18-50; be able to read and write at an intermediate level (Education > 8 years or more); social anxiety scores above 34 for the SIAS, above 19 for the SPIN and above 20 for the BSPS; and the the presence of observable clinical symptoms supporting the diagnosis of a social anxiety disorder on Axis I.

Exclusion Criteria:

* Diagnosis of affective psychosis; currently clinically stable [score of 3 or less of the SAPS ratings; Global Assessment Scale score (Endicott, et al., 1976) of ≥ 50]; have no significant presence of social anxiety (score on scales below cut-off); hospitalized or hospitalized at the time of recruitment; and a change medication within the past 6 weeks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Social anxiety symptom reduction | 13-week intervention program
  To compare the effectiveness in social anxiety symptom reduction of a 13-week group CBT for social anxiety adapted for people with schizophrenia relative to a control condition involving participants who will be receiving standard care only, followed by the proposed intervention on a wait-list basis

SECONDARY OUTCOMES:
Positive and negative symptoms of schizophrenia reduction | 13-week intervention program
  To measure the effect of a group CBT intervention for social anxiety on positive and negative symptoms of schizophrenia.

CONTACTS AND LOCATIONS:
Locations (1):
- RUIS McGill CBT Teaching & Research Program, Montreal, Quebec, Canada